CLINICAL TRIAL: NCT02398604
Title: Allogeneic Human MEsenchymal Stem Cell (hMSC) Injection in Patients With Hypoplastic Left Heart Syndrome: An Open Label Pilot Study.
Brief Title: Allogeneic hMSC Injection in Patients With Hypoplastic Left Heart Syndrome
Acronym: ELPIS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was closed due to Sponsor switched to Longeveron. New Identifier is NTC03525418
Sponsor: Longeveron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140718
Record Dates: First submitted 2014-12-24; First posted 2015-03-25 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Pediatrics; HLHS
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Intervention Model Description: 20 patients and 10 patients will be controls with a total of 30 HLHS patients.
Masking Description: HLHS patients which will be randomized to the treatment and control arms in a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A - Allo-hMSCs (Experimental): Group A: Fifteen (20) patients will be treated with Allogenic human mesenchymal stem cells (Allo-hMSCs): A concentration of 5 million cells/ml delivered in a dose of 2.5 x 10^5 cells per kg of recipient (5 million/20kg) Allo-hMSCs. The entire dose of the cells will be divided and delivered in 6-10 open intramyocardial injections during the BDCPA operation.
  Interventions: Drug: Allo-hMSCs
- Group B (Placebo Comparator): Group B: Fifteen (10) patients will be treated with a placebo comparator. The placebo will be divided and delivered in 6-10 open intramyocardial injections during the BDCPA operation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allo-hMSCs — Allogeneic Human Mesenchymal Stem Cells
  Other Names: stem cells; Allogeneic Human Mesenchymal Stem Cells
  Arms: Group A - Allo-hMSCs
Drug: Placebo — Placebo
  Other Names: Placebo comparator
  Arms: Group B

SUMMARY:
This study is intended to evaluate the safety and feasibility of intramyocardial injection of allogeneic mesenchymal cells during the Bi-Directional Cavopulmonary Anastomosis (BDCPA) surgery for hypoplastic left heart syndrome (HLHS) pediatric patients.

DETAILED DESCRIPTION:
This is an open label study, intended as a safety and efficacy assessment prior to a full comparator study. In this Phase I study, cells administered will be delivered in 6-10 intramyocardial injections that will be tested in 20 patients and 10 patients will be controls with a total of 30 HLHS patients.

A total of 30 patients with HLHS will be enrolled in a staged enrollment process. In this open-labeled study, a maximum of 20 patients will eventually receive intramyocardial injection of the allogeneic mesenchymal stem cells and 10 control patients with no cell injection. The enrollment of the patients will occur in two stages groups: Group A and Group B. In Group A, 10 consecutive HLHS patients will be initially enrolled in the allogenic MSCs treatment arm to determine feasibility and safety. After 6 months of the last enrolled patient in Group A, all Group A patients will be assessed in order to determine whether it is feasible and safe, including the harvesting, processing, and administering of the allogeneic MSCs. Thereafter, Group B will start enrolling a total of 20 HLHS patients which will be randomized to the treatment and control arms in a 1:1 ratio, respectively, in order to have 10 allogeneic MSCs-treated patient and 10 control patients. At the completion of this Phase I clinical study, the total enrolled cohort will be 20 patients treated with allogeneic MSCs and 10 patients in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hypoplastic left heart syndrome (all types) requiring BDCPA surgery.

Exclusion Criteria:

* Have HLHS and restrictive or intact atrial septum.
* Be undergoing the Norwood procedure that do not have HLHS.
* Have significant coronary artery sinusoids.
* Require mechanical circulatory support prior to surgery.
* Have an underlying evidence of arrhythmia requiring anti-arrhythmia therapy.
* Parent or guardian unwilling or unable to comply with necessary follow-up(s)
* Be serum positive for HIV, hepatitis BsAg (B Surface Antigen) or viremic hepatitis C.
* Be unsuitable for inclusion in the study, in the opinion of the investigator.
* Need for concomitant surgery for aortic coarctation or tricuspid valve repair.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2015-04; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Monitor major adverse cardiac events | 1 month after injection
  Monitoring of events includes death, sustained/symptomatic ventricular tachycardia requiring intervention with inotropic support, aggravation of heart failure, new myocardial infarction, unplanned cardiovascular operation for cardiac tamponade and infection in the first month after injection, and serially afterwards.

SECONDARY OUTCOMES:
Composite Change from baseline in right ventricular function, right ventricular end-diastolic volume, right ventricular end-systolic volume, right ventricular end-systolic diameter and tricuspid regurgitation | baseline, 24 weeks and 1 year
  as measured by serial echocardiograms and MRI scans.
Number of participants with incidence of mortality or need for transplantation after the BDCPA operation | One year after injections
  Assessed through the number of participants with adverse events, hospitalizations, or transplantations.
Composite Changes in somatic growth velocity over time (weight, height, head circumference) from the BDCPA operation | 12 months post operative
  Changes in weight, height, and head circumference will be measured
Assessment of Co-morbidity | up to 12 months follow-up
  Assessment of cardiovascular mortality, all-cause morbidity, Cardiovascular morbidity, re-hospitalizations, need for transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Oliva, MD, Principal Investigator — Longeveron Inc.
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Interdisciplinary Stem Cell Institute — http://isci.med.miami.edu